CLINICAL TRIAL: NCT00430625
Title: A Multicenter, Randomized, Double-Blind, Parallel Group, Two-Dose Study of Gene-Activated® Human Glucocerebrosidase (GA-GCB) Enzyme Replacement Therapy in Patients With Type 1 Gaucher Disease
Brief Title: A Study of Gene-Activated® Human Glucocerebrosidase (GA-GCB) Enzyme Replacement Therapy in Gaucher Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TKT032
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Results first posted 2010-09-10 (Estimated); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Gaucher Disease, Type 1
Keywords: VPRIV®; Enzyme Replacement Therapy; Gaucher disease; glucocerebrosidase; beta-glucocerebrosidase; Acid beta-glucocerebrosidase; glucosylceramidase; D-glucosyl-N-acylsphingosine glucohydrolase; gene activation; human
MeSH Terms: conditions — Gaucher Disease | interventions — Glucosylceramidase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VPRIV®-45 U/kg, IV, every other week (Experimental): VPRIV® (velaglucerase alfa, Gene Activated® human glucocerebrosidase, GA-GCB)
  Interventions: Biological: VPRIV ®,
- VPRIV®-60 U/kg, IV, every other week (Experimental): VPRIV® (velaglucerase alfa, Gene Activated® human glucocerebrosidase,GA-GCB)
  Interventions: Biological: VPRIV ®,

INTERVENTIONS:
Biological: VPRIV ®, — Intravenous (IV) infusion, every other week via intravenous infusion for 12 months
  Other Names: VPRIV®; velaglucerase alfa; GA-GCB; Gene-activated® human glucocerebrosidase

SUMMARY:
Gaucher disease is a rare lysosomal storage disorder caused by the deficiency of the enzyme glucocerebrosidase (GCB). Due to this deficiency of functional GCB, glucocerebroside accumulates within macrophages leading to cellular engorgement, organomegaly, and organ system dysfunction. The purpose of this study is to evaluate the efficacy of every other week dosing of Gene-Activated® Human Glucocerebrosidase (GA-GCB, velaglucerase alfa) at doses of 45 and 60 U/kg in treatment-naïve patients with type 1 Gaucher disease.

DETAILED DESCRIPTION:
Type 1 Gaucher disease, the most common form, accounts for more than 90% of all cases and does not involve the Central Nervous System (CNS). Typical manifestations of type 1 Gaucher disease include hepatomegaly, splenomegaly, thrombocytopenia, bleeding tendencies, anemia, hypermetabolism, skeletal pathology, growth retardation, pulmonary disease, and decreased quality of life. Gene-Activated® human glucocerebrosidase (GA-GCB; velaglucerase alfa) is produced in a continuous human cell line using proprietary gene-activation technology and has an identical amino acid sequence to the naturally occurring human enzyme. Velaglucerase alfa contains terminal mannose residues that target the enzyme to the macrophages-the primary target cells in Gaucher disease. This study was designed to determine the efficacy, safety and pharmacokinetics of GA-GCB in men, women, and children with Type 1 Gaucher disease. Each patients duration of treatment was 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a documented diagnosis of type 1 Gaucher disease, as determined by deficient glucocerebrosidase (GCB) activity relative to normal as measured in leukocytes or by genotype analysis and is willing and able to provide written informed consent prior to initiating any study-related procedures
* Patient is at least 2 years of age
* Patient has Gaucher disease-related anemia and
* Patient has at least moderate splenomegaly or
* Patient has Gaucher disease-related thrombocytopenia or
* Patient has a readily palpable enlarged liver
* Patient has not received treatment for Gaucher disease within 30 months prior to study entry
* Female patients of child-bearing potential agree to use a medically acceptable method of contraception. Male patients must agree to use a medically acceptable method of birth control.
* Patient must be sufficiently cooperative to participate in the study as judged by the Investigator.

Exclusion Criteria:

Includes:

* Patient has type 2 or 3 Gaucher disease or is suspected of having type 3 Gaucher disease
* Patient is antibody-positive to imiglucerase during screening or has experienced an anaphylactic reaction to imiglucerase
* Patient has received treatment with any investigational drug or device within the 30 days prior to study entry
* Patient is Human immunodeficiency virus (HIV) positive
* Patient is hepatitis positive
* Patient presents with iron, folic acid and/or vitamin B12 deficiency sustained anemia during screening
* Patient, patient's parent(s), or patient's legal guardian(s) is/are unable to understand the nature, scope, and possible consequences of the study
* Patient has a significant comorbidity(ies)that might affect study data or confound the study results
* Patient is a pregnant and/or lactating female
* Patient is unable to comply with the protocol or is unlikely to complete the study, as determined by the Investigator

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-02-15 (Actual); Primary Completion 2009-04-01 (Actual); Study Completion 2009-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- Hipolito Yrigoyen, Buenos Aires, Argentina
- Shaare Zedek Medical Center, Jerusalem, Israel
- Sociedad Espanola de Socorros Mutuos, Asunción, Paraguay
- National Research Center for Haematology, Moscow, Russia
- La Rabta Hospital, Tunis, Tunisia

REFERENCES:
- [Derived] Zimran A, Elstein D, Gonzalez DE, Lukina EA, Qin Y, Dinh Q, Turkia HB. Treatment-naive Gaucher disease patients achieve therapeutic goals and normalization with velaglucerase alfa by 4years in phase 3 trials. Blood Cells Mol Dis. 2018 Feb;68:153-159. doi: 10.1016/j.bcmd.2016.10.007. Epub 2016 Oct 21. PMID 27839979
- See also: Shire product Information web site — http://www.vpriv.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Type 1 Gaucher disease patients (pts) >2 years. The first patient (pt) was enrolled in the study on 15 February 2007.
Pre-assignment Details: Gaucher disease-related anemia and at least 1 of the following: moderate splenomegaly, thrombocytopenia or palpable enlarged liver. Patients were not to have received any treatment for Gaucher disease within 30 months of study entry. Patients randomized to receive VPRIV®(45 or 60 U/kg)every other week by intravenous (IV) infusion.
Groups:
- VPRIV® (45 U/kg, IV, Every Other Week); VPRIV® (60 U/kg, IV, Every Other Week): velaglucerase alfa, Gene Activated® human glucocerebrosidase, GA-GCB
Period: Overall Study
Arm/Group | VPRIV® (45 U/kg, IV, Every Other Week) | VPRIV® (60 U/kg, IV, Every Other Week)
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VPRIV® (45 U/kg, IV, Every Other Week) | VPRIV® (60 U/kg, IV, Every Other Week) | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 4 | 7
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 30.0 (16.75) [6 to 62] | 23.5 (11.77) [4 to 42] | 25 (15.28) [4 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 8 | 7 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  Paraguay | 6 | 5 | 11
  Argentina | 1 | 0 | 1
  Russian Federation | 3 | 0 | 3
  Israel | 1 | 6 | 7
  Tunisia | 2 | 1 | 3
Baseline Spleen volume [Median (Full Range); unit: Percent of body weight] — Normal spleen volume is defined as 0.2 percentage of body weight.
  Percent of body weight | 2.9 [0.5 to 13.0] | 2.8 [0.4 to 7.4] | 2.9 [0.4 to 13.0]
Baseline hemoglobin concentration per treatment group [Median (Full Range); unit: g/dL] — Modified baseline used for analysis (defined as average of screening and baseline values)
  g/dL | 10.90 (1.278) [8.45 to 12.85] | 10.83 (1.272) [7.05 to 12.25] | 10.85 (1.248) [7.05 to 12.85]
Baseline liver volume [Median (Full Range); unit: Percent of body weight] — Normal liver volume is defined as 2.5 percent of body weight.
  Percent of body weight | 3.50 [2.3 to 7.2] | 3.65 [2.4 to 8.0] | 3.5 [2.3 to 8.0]
Baseline platelet counts per treatment group [Median (Full Range); unit: (x10^9/L)] — Modified baseline used for analysis (defined as average of screening and baseline values)
  (x10^9/L) | 58.00 (59.56) [13 to 264] | 66.75 (111.91) [47 to 438] | 65.5 (86.71) [13 to 438]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 12 Months in Hemoglobin Concentration for the 60 U/kg Treatment Group.
Description: Efficacy endpoint
Time Frame: Week 53
Population: 12 patients in the 60 U/kg group were analyzed for efficacy in the intent to treat (ITT) population.
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | VPRIV® (60 U/kg, IV, Every Other Week)
Number analyzed (Participants) | 12
g/dL | 2.429 [1.717 to 3.141]
Statistical Analysis 1: Comparison: VPRIV® (60 U/kg, IV, Every Other Week); Primary endpoint was based solely on the 60 U/kg treatment arm; Test type: Superiority or Other; p < 0.0001, paired t-test; Mean Difference (Final Values) = 2.429, 95% CI 2-sided [1.717 to 3.141], Standard Error of Mean 0.324

2. Secondary Outcome: Change From Baseline to 12 Months in Hemoglobin Concentration in 45 U/kg Treatment Group
Time Frame: Week 53
Population: 13 patients in the 45 U/kg group were analyzed for efficacy in the intent to treat (ITT) population.
Measure: Mean (95% Confidence Interval); unit: (g/dL)
Arm/Group | VPRIV® (45 U/kg, IV, Every Other Week)
Number analyzed (Participants) | 13
(g/dL) | 2.438 [1.488 to 3.389]

3. Secondary Outcome: Change From Baseline to 12 Months in Platelet Counts for Each Treatment Group.
Description: intent to treat (ITT) Population
Time Frame: Week 53
Population: 12 patients in the 60 U/kg group and 13 patients in the 45 U/kg group were analyzed for efficacy in the intent to treat (ITT) population.
Measure: Mean (95% Confidence Interval); unit: x10^9/L
Arm/Group | VPRIV® (45 U/kg, IV, Every Other Week) | VPRIV® (60 U/kg, IV, Every Other Week)
Number analyzed (Participants) | 13 | 12
x10^9/L | 40.92 [11.20 to 70.64] | 50.88 [23.97 to 77.78]

4. Secondary Outcome: Change From Baseline to 12 Months in Normalized Liver Volume (Percent Body Weight) for Each Treatment Group (Measured by Magnetic Resonance Imaging (MRI)
Description: Liver Volume has been normalized for percentage of body weight for each treatment arm. Liver size relative to body weight = (Liver volume [cc]/Body weight [kg])*100
Time Frame: Week 51
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Percent body weight
Arm/Group | VPRIV® (45 U/kg, IV, Every Other Week) | VPRIV® (60 U/kg, IV, Every Other Week)
Number analyzed (Participants) | 13 | 12
Percent body weight | -0.30 [-0.92 to 0.32] | -0.84 [-1.58 to -0.11]

5. Secondary Outcome: Change From Baseline to 12 Months in Normalized Spleen Volume (Percent Body Weight) for Each Treatment Group (Measured by Magnetic Resonance Imaging (MRI))
Description: 12 patients in the 60 U/kg group and 13 patients in the 45 U/kg group were analyzed for efficacy in the intent to treat (ITT) population. Spleen Volume has been normalized for percent of body weight for each treatment arm. Spleen size relative to body weight = (Spleen volume [cc]/Body weight [kg])*100
Time Frame: Week 51
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Percent body weight
Arm/Group | VPRIV® (45 U/kg, IV, Every Other Week) | VPRIV® (60 U/kg, IV, Every Other Week)
Number analyzed (Participants) | 13 | 12
Percent body weight | -1.87 [-3.17 to -0.57] | -1.92 [-3.04 to -0.79]

6. Secondary Outcome: Percent Change From Baseline to 12 Months in Plasma Chitotriosidase for Each Treatment Group
Description: Percent Change from Baseline to Weeks 53 by Randomized velaglucerase alfa Treatment Group - Subset of intent to treat (ITT) Population who were wild type homozygous for chitotriosidase.
Time Frame: Week 53
Population: 2 patients in the 60 U/kg group and 7 patients in the 45 U/kg group who were wild type for the chitotriosidase mutation were analyzed; remaining patients were deficient in chitotriosidase activity.
Measure: Number; unit: Percent
Arm/Group | VPRIV® (45 U/kg, IV, Every Other Week) | VPRIV® (60 U/kg, IV, Every Other Week)
Number analyzed (Participants) | 2 | 7
Percent | -61.16 (7.768) | -69.65 (17.65)

7. Secondary Outcome: Percent Change From Baseline to 12 Months in Chemokine (C-C Motif) Ligand 18 (CCL18)
Time Frame: Week 53
Population: 12 patients in the 60 U/kg group and 13 patients in the 45 U/kg group were analyzed.
Measure: Number; unit: Percent
Arm/Group | VPRIV® (45 U/kg, IV, Every Other Week) | VPRIV® (60 U/kg, IV, Every Other Week)
Number analyzed (Participants) | 13 | 12
Percent | -46.76 (7.623) | -66.02 (5.358)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored either from time of informed consent/assent (Amendment 1) or from the first infusion (original protocol) through 30 days after the last infusion (Week 53).
Description: Adverse events may have been discovered through observation/examination of the patient, questioning of the patient or complaint by the patient. Adverse Events could have included unexpected laboratory values that became significantly out of range. Other adverse events were determined to be possibly/probably related to VPRIV by the Investigator.
Arm/Group | VPRIV® (45 U/kg, IV, Every Other Week) | VPRIV® (60 U/kg, IV, Every Other Week)
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/12
Other Adverse Events (participants affected / at risk) | 9/13 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VPRIV® (45 U/kg, IV, Every Other Week) (N=13) | VPRIV® (60 U/kg, IV, Every Other Week) (N=12)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 1 (1) — Considered not related by investigator.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VPRIV® (45 U/kg, IV, Every Other Week) (N=13) | VPRIV® (60 U/kg, IV, Every Other Week) (N=12)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hyperproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to small sample sizes no conclusions could be drawn on Quality of life (QOL).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Shire's agreements with investigators vary. All agreements provide Shire the right to embargo communications regarding trial results prior to public release for a period ≤180 days from the time submitted to Shire for review. Shire does not prohibit publication, but can require the removal of confidential information (excluding trial results) and can request postponement of a single-center publication until after disclosure of the trial's multi-center publication.